CLINICAL TRIAL: NCT03364725
Title: Toward Elimination of Hepatitis C Virus (HCV): A Pilot Study Combining HCV and Addiction Treatment of Young Suburban Heroin Users (SHU) That Addresses Barriers to Care
Brief Title: Toward Elimination of Hepatitis C Virus (HCV): A Pilot Study
Acronym: ELIMINATEC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Id Care (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Ronald Nahass, Principle Invesigator, Id Care
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIS # 11-507
Record Dates: First submitted 2017-12-01; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Hepatitis C; Addict Heroin
MeSH Terms: conditions — Hepatitis C | interventions — glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label Treatment Arm (Experimental): Treatment arm using Glecaprevir-pibrentasvir for treatment of all patients
  Interventions: Drug: Glecaprevir-pibrentasvir

INTERVENTIONS:
Drug: Glecaprevir-pibrentasvir — Glecaprevir-pibrentasvir will be dispensed to 30 patients recently detoxed off heroin in an acute detox center.

SUMMARY:
To demonstrate that colocation treatment of substance use disorder and Hepatitis C infection concurrently while proving addiction counselling will achieve increased duration of sobriety and elimination of Hepatitis C virus in study participants.

DETAILED DESCRIPTION:
To demonstrate that colocation treatment of substance use disorder and Hepatitis C infection concurrently while proving addiction counselling will achieve increased duration of sobriety and elimination of Hepatitis C virus in study participants.

Primary objective:

1. Cure rates (SVR-12, HCV plasma RNA not quantifiable 12 weeks after last dose of treatment) of HCV in 30 recently identified PWIDS under 30 years old

Secondary objectives:

1. Rate of sobriety maintenance for 1 year after enrollment
2. Re-infection rate with HCV over 1 year after enrollment
3. Re-admission rates for detox
4. Cravings

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 30
* Successfully detoxed at PHBH from opioids
* Agree to participate in a closely monitored program
* Positive HCV VL > 5,000 on two tests
* Minimum one follow-up visit after discharge from PHBH to be enrolled
* Any genotype
* APRI less than 1 and Fibrosure less than 0.45
* Negative pregnancy test in women and females must agree to acceptable contraception during treatment of HCV. Oral contraceptives that do not contain ethinyl estradiol are allowed with Mavyret
* Treatment naïve for HCV
* Signed informed consent

Exclusion Criteria:

* Cirrhosis
* Co-infection with HIV or HBV
* Inability to comply with treatment or follow up
* Renal failure with GFR less than 50 mL/min5*
* Any prior treatment for HCV
* Diabetes with HgA1c more than 8.0
* Clinically significant abnormalities, other than HCV infection, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead electrocardiogram (ECG) that make the subject an unsuitable candidate for this study in the opinion of the investigator, including, but not limited to:

  * ALT/AST > 10x normal value,
  * WBC with ANC < 1500 cell/ul,
  * Hemoglobin < LLN,
  * Treatment for cancer or lymphoma in the past 5 years,
  * Hemoglobin A 1C > 8%.
* Any uncontrolled psychiatric, cardiac, respiratory, gastrointestinal, hematologic, neurologic, psychiatric, or other medical disease or disorder, which is unrelated to the existing HCV infection which in the opinion of the PI would prevent adherence to and participation in the trial.
* Hypersensitivity to naltrexone or polylactide-co-glycolide (PLG) microspheres

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-15 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Cure rate of Hepatitis C Infection | 12 weeks after treatment completion viral load measure
  Cure rates (SVR-12, HCV plasma RNA not quantifiable 12 weeks after last dose of treatment) of HCV in 30 recently identified PWIDS under 30 years

SECONDARY OUTCOMES:
Sobriety from Drug Use | 1 year
  Rate of sobriety maintenance for 1 year after enrollment
Hepatitis C Reinfection Rate | 1 year
  Re-infection rate with HCV over 1 year after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Nahass, MD, Principal Investigator — Id Care
Locations (1):
- ID CARE, Hillsborough, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No